CLINICAL TRIAL: NCT00245206
Title: Metabolic Effects of Newer Antipsychotics in Older Patients
Brief Title: Side Effects of Newer Antipsychotics in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dilip V. Jeste, Psychiatry, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH071536 (NIH); DATR A5-ETSE (Registry Identifier: Clinicaltrials.gov); R01MH071536 (NIH)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Schizophrenia; Alzheimer's Disease; Dementia
Keywords: Antipsychotic; Diabetes; Hyperlipidemia; Stroke
MeSH Terms: conditions — Schizophrenia; Alzheimer Disease; Dementia; Diabetes Mellitus; Hyperlipidemias; Stroke | interventions — Aripiprazole; Olanzapine; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: Risperdal (Experimental): Participants randomized to this arm will be prescribed risperdal. They will continue to be followed by their psychiatrist. In addition, they will take part in ongoing biological, cognitive, and psycho-social assessments with study staff.
  Interventions: Drug: Risperidone
- 3: Aripiprazole (Experimental): Participants randomized to this arm will be prescribed aripiprazole. They will continue to be followed by their psychiatrist. In addition, they will take part in ongoing biological, cognitive, and psycho-social assessments with study staff.
  Interventions: Drug: Aripiprazole
- 4: Olanzapine (Experimental): Participants randomized to this arm will be prescribed olanzapine. They will continue to be followed by their psychiatrist. In addition, they will take part in ongoing biological, cognitive, and psycho-social assessments with study staff.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Aripiprazole — Participant will take aripiprazole. Dosing will be determined by each participant's psychiatrist.
  Arms: 3: Aripiprazole
Drug: Olanzapine — Participant will take olanzapine. Dosing will be determined by each participant's psychiatrist.
  Arms: 4: Olanzapine
Drug: Risperidone — Participant will take risperidone. Dosing will be determined by each participant's psychiatrist.
  Other Names: Risperidal
  Arms: 1: Risperdal

SUMMARY:
This study will compare four atypical antipsychotic medications in terms of the risk of specific side effects each of them presents in middle-aged and elderly individuals.

DETAILED DESCRIPTION:
Atypical antipsychotic medications introduced within the last decade have been used increasingly for the treatment of several types of psychotic disorders and severe behavioral disturbances in older individuals. This trend is primarily due to a decrease in side effects caused by the new medications, as compared to conventional neuroleptic medications. There is a lower risk for developing tardive dyskinesia and extrapyramidal symptoms, both of which are movement abnormalities, with new antipsychotic medications. However, there has been a growing concern that the newer medications can cause a different set of potentially serious adverse side effects. Specifically, they may cause long-term metabolic, cardiovascular, and cerebrovascular effects, which may result in weight gain, diabetes, or stroke. This study will compare four atypical antipsychotic medications in terms of the risk of metabolic, cardiovascular, and cerebrovascular side effects that each presents in middle-aged and elderly individuals.

Participants in this open-label study will be randomly assigned to receive one of three atypical antipsychotic medications: aripiprazole; olanzapine; or risperidone. Although assignment is random, a technique that may reflect the participant's own interests or the researcher's knowledge of relevant participant characteristics will be used to assign the participant to a medication. Dosing will be determined by each participant's psychiatrist. Participants will be followed for up to 5 years to assess the side effects of the study medications, with study visits at baseline, Week 6, and every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of a disease or disorder that requires treatment with an atypical antipsychotic medication

Exclusion Criteria:

* N/A

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2005-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Measured at baseline, Week 6, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
  Change in body mass index (BMI) between each study visit. weight and height will be combined to report BMI in kg/m^2. (This hypothesis is non-directional because of uncertainties with respect to significant between-drug differences on these measures.)
Change in Fasting Plasma Glucose (FPG) | Measured at baseline, Week 6, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
  Blood sample collected to measure Fasting Plasma Glucose (FPG) to determine if there are changes between study visits. (This hypothesis is non-directional because of uncertainties with respect to significant between-drug differences on these measures.)
Change in LDL cholesterol, HDL cholesterol, and triglycerides | Measured at baseline, Week 6, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
  Lipid Panel collected to measure LDL cholesterol, HDL cholesterol, and triglycerides and determine if there are changes between study visits. (This hypothesis is non-directional because of uncertainties with respect to significant between-drug differences on these measures.)

CONTACTS AND LOCATIONS:
Overall Officials: Dilip V. Jeste, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin H, Shih PA, Golshan S, Mudaliar S, Henry R, Glorioso DK, Arndt S, Kraemer HC, Jeste DV. Comparison of longer-term safety and effectiveness of 4 atypical antipsychotics in patients over age 40: a trial using equipoise-stratified randomization. J Clin Psychiatry. 2013 Jan;74(1):10-8. doi: 10.4088/JCP.12m08001. Epub 2012 Nov 27. PMID 23218100
- [Derived] Jin H, Meyer J, Mudaliar S, Henry R, Khandrika S, Glorioso DK, Kraemer H, Jeste D. Use of clinical markers to identify metabolic syndrome in antipsychotic-treated patients. J Clin Psychiatry. 2010 Oct;71(10):1273-8. doi: 10.4088/JCP.09m05414yel. PMID 21062616